CLINICAL TRIAL: NCT02165748
Title: Severe Intraoperative Hyperglycemia During Craniotomy and Postoperative Infections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Federico Bilotta, Dr, University of Roma La Sapienza
Other Study IDs: IntraopHypegl&Infections
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Patients Undergoing Craniotomy for Brain Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Aim of this prospective observational study -in patients undergoing craniotomy for supra or infratentorial surgery as elective or emergency procedure- is to test the hypothesis that severe intraoperative hyperglycemia (BGC ≥180mg/dl) is associated with an increased incidence of infections within the first postoperative week (pneumonia, blood stream, urinary, surgical site/wound and cerebral infections)(NCT01923571).

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Undergoing elective or emergency craniototmy

Exclusion Criteria:

* Age <18

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing craniotomy for brain surgery
Sampling Method: Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of infections in patients presenting intraoperative severe hyperglycemia during craniotomy | 7 days

SECONDARY OUTCOMES:
survival during the study period | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Federico Bilotta, MD, PhD, Principal Investigator — Department of Anesthesiology, University of ROme "La Sapienza"
Locations (1):
- University of ROme "La Sapienza", Rome, Italy

REFERENCES:
- [Derived] Gruenbaum SE, Toscani L, Fomberstein KM, Ruskin KJ, Dai F, Qeva E, Rosa G, Meng L, Bilotta F. Severe Intraoperative Hyperglycemia Is Independently Associated With Postoperative Composite Infection After Craniotomy: An Observational Study. Anesth Analg. 2017 Aug;125(2):556-561. doi: 10.1213/ANE.0000000000001946. PMID 28181933